CLINICAL TRIAL: NCT01237379
Title: Peroxisomal Defects and Familial Risk for Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Robert McNamara, Associate Professor, University of Cincinnati
Other Study IDs: McNamara NARSAD
Record Dates: First submitted 2010-10-21; First posted 2010-11-09 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Bipolar Disorder; Mania
MeSH Terms: conditions — Bipolar Disorder; Mania

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Laboratory methods: The gas chromatography procedure used to determine red blood cell fatty acid composition. Briefly, total fatty acid composition will be determined. Indices of peroxisome function, including (1) plasma very long chain fatty acids concentrations, (2) plasma bile acid C27 intermediate concentrations, (3) plasma pipecolic acid concentrations, and (4) RBC plasmalogen concentrations, will be determined by liquid chromatography tandem mass spectrometry and gas chromatography. Plasma cytokine and C-Reactive Protein (CRP)concentrations will be determined. All blood analyses will be performed by a technician blinded to diagnostic group identity.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Health Controls
- Bipolar Patients with High-Risk of Mania
- Bipolar Patients with Ultra-High Risk
- First Manic Episode Bipolar Youth

SUMMARY:
The purpose of this study is to screen for peroxisome defects in child and adolescent offspring of Bipolar Disorder I (BD-I) parents at different stages of risk for transitioning to mania and following the onset of mania.

Prediction 1: Youth with an elevated risk for developing BD-I and first-episode manic patients will exhibit graded deficits in measures of peroxisomal function compared with healthy controls.

Prediction 2: Indices of peroxisomal function will be correlated with Red Blood Cells Docosahexaenoic acid (DHA) composition.

Prediction 3: Graded deficits in measures of peroxisomal function will be inversely correlated with manic and depression symptom severity scores.

DETAILED DESCRIPTION:
Overall Study Design: This study entails collecting fasting venous blood (20 ml) from, and administering the 'omega-3 questionnaire' to, subjects being recruited from ongoing National Institute of Mental Health (NIMH)-sponsored trials within the Department of Psychiatry, University of Cincinnati College of Medicine. Specifically, blood will be collected from 20 healthy controls (i.e., no personal or family history of any Axis I mood disorder according to the Diagnostic and Statistical Manual of Mental Disorders-IV [DSM-IV]) and 20 asymptomatic high-risk (i.e., have a biological parent with BD-I) adolescents (aged 10-18 years old) recruited for study MH077138 (UC-IRB #: 07-04-10-03, BITREC Project 3; PI: DelBello), 20 ultra-high risk (i.e., have a biological parent with BD-I and a Major Depressive Disorder (MDD) diagnosis) recruited for study MH083924 (UC-IRB #: 04-09-15-03, CO-Principal Investigators DelBello/McNamara), and 20 adolescents who are admitted for their first hospitalization and who have a diagnosis of BD-I recruited for study MH080973 (UC-IRB #: 08-10-30-01, Principal Investigator: DelBello). Blood will then be processed, and de-identified tubes sent to the Kennedy Krieger Institute, Peroxisomal Diseases Section, to determine the following measures of peroxisomal function: (1) plasma very long chain fatty acids (C24:0 & C26:0) concentrations, (2) plasma bile acid C27 intermediate (dehydrocrepenynic acid {DHCA},tetrahydrocannabinolic acid {THCA})concentrations, (3) plasma pipecolic acid concentrations, and (4) Red Blood Cell (RBC) plasmalogen concentrations. Additionally, RBC fatty acid composition will be determined by gas chromatography, and platelet function and plasma inflammatory markers assayed using commercially available kits according to manufacturer's instructions.

ELIGIBILITY:
Subject characteristics: All subjects will be 10-18 year old males and females. Up to 80 patients will be enrolled in this study. Subjects will be screened according to previously approved individual study criteria (UC-IRB #: 07-04-10-03; 04-09-15-03; 08-10-30-01).

Inclusion Criteria:

* 10 -18 year old males & females
* Based on currently enrolled study.

Exclusion Criteria:

* Based on currently enrolled study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects: In order to accomplish this aim, 20 healthy controls, 20 high-risk, 20 ultra-high risk, and 20 first-episode manic youth (ages 10-18 years old) will be recruited at a rate of 1 subject/group per month over the first 20 months. Subjects being recruited from the following IRB approved NIMH-sponsored trials: MH077138 (UC-IRB #: 07-04-10-03, BITREC Project 3; PI: DelBello), MH083924 (UC-IRB #: 04-09-15-03, CO-PIs DelBello/McNamara), and MH080973 (UC-IRB #: 08-10-30-01, PI: DelBello).
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Youth with an elevated risk for developing BD-I and first-episode manic patients will exhibit graded deficits in measures of peroxisomal function compared with healthy controls. | 1 day
  Prediction 1: Youth with an elevated risk for developing BD-I and first-episode manic patients will exhibit graded deficits in measures of peroxisomal function compared with healthy controls.

SECONDARY OUTCOMES:
peroxisomal function will be inversely correlated with manic and depression symptom severity scores. | 1 day
  Prediction 3: Graded deficits in measures of peroxisomal function will be inversely correlated with manic and depression symptom severity scores.
Indices of peroxisomal function will be correlated with RBC DHA composition. | 1 day
  Prediction 2: Indices of peroxisomal function will be correlated with RBC DHA composition.

CONTACTS AND LOCATIONS:
Overall Officials: Robert McNamara, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States